CLINICAL TRIAL: NCT07018258
Title: Optimal Patient Positioning for Erector Spinae Plane Block: Effects on Postoperative Analgesia and Patient Satisfaction"
Brief Title: Optimal Patient Positioning for Erector Spinae Plane Block in Laparoscopic Cholecystectomy:
Acronym: ESP-POSTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Veli Fahri Pehlivan, Assistant Professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cevher
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Laparoscopic Cholecystectomy; Anesthesia, Regional; Pain Management
Keywords: Erector Spinae Plane Block; Patient Positioning; Ultrasound-Guided Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Parapsychology; Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive ESP block in either the lateral, prone, or sitting position prior to laparoscopic cholecystectomy.
Who Masked: Outcomes Assessor
Masking Description: The person evaluating postoperative pain scores and satisfaction will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lateral Position Group (Experimental): Patients in this group will receive bilateral erector spinae plane (ESP) block at the T7 level in the lateral decubitus position under ultrasound guidance before laparoscopic cholecystectomy.
  Interventions: Procedure: Erector Spinae Plane (ESP) Block
- Prone Position Group (Experimental): Patients in this group will receive bilateral erector spinae plane (ESP) block at the T7 level in the lateral decubitus position under ultrasound guidance before laparoscopic cholecystectomy.
  Interventions: Procedure: Erector Spinae Plane (ESP) Block
- Sitting Position Group (Experimental): Patients in this group will receive bilateral erector spinae plane (ESP) block at the T7 level in the lateral decubitus position under ultrasound guidance before laparoscopic cholecystectomy.
  Interventions: Procedure: Erector Spinae Plane (ESP) Block

INTERVENTIONS:
Procedure: Erector Spinae Plane (ESP) Block — Ultrasound-guided bilateral erector spinae plane (ESP) block performed at the T7 vertebral level. The intervention will be applied in three different patient positions-lateral, prone, or sitting-prior to laparoscopic cholecystectomy.
  Other Names: Ultrasound-guided ESP block

SUMMARY:
This randomized clinical study aims to compare the postoperative analgesic efficacy, analgesic consumption, and patient satisfaction of erector spinae plane (ESP) block administered in three different patient positions-lateral, prone, and sitting-in individuals undergoing elective laparoscopic cholecystectomy. The study also evaluates the variation in skin-to-block site distance depending on patient positioning.

DETAILED DESCRIPTION:
Erector spinae plane (ESP) block is a relatively recent regional anesthesia technique performed under ultrasound guidance, widely used for managing acute postoperative pain. While the ESP block is known for its safety, simplicity, and versatility, there is limited evidence regarding the influence of patient positioning on its clinical effectiveness and technical performance.

This prospective, randomized, single-blind study investigates the impact of administering bilateral ESP block at the T7 vertebral level in three different patient positions: lateral decubitus, prone, and sitting. The study includes adult patients (aged 18-65, ASA I-II) undergoing elective laparoscopic cholecystectomy under general anesthesia.

Primary outcomes include postoperative pain scores (VAS and NRS). Secondary outcomes include total rescue analgesic consumption (tramadol), time to first analgesic requirement, patient satisfaction scores (Likert scale), and measurement of the skin-to-block site distance across different positions. Data will be collected at defined intervals up to 24 hours postoperatively.

The findings are expected to inform clinicians on the optimal patient positioning for ESP block to enhance block efficacy and patient comfort during laparoscopic abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Scheduled for elective laparoscopic cholecystectomy
* ASA physical status I-II
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Allergy to local anesthetics
* History of chronic opioid use or substance abuse
* Coagulopathy or current anticoagulant therapy
* Local infection at the block site
* Severe spinal deformities or scoliosis
* BMI > 35 kg/m²
* Pregnancy or breastfeeding
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score (VAS) | 0, 2, 4, 6, 12, and 24 hours postoperatively
  Pain intensity will be assessed using the Visual Analog Scale (VAS, 0-10) at multiple time points following laparoscopic cholecystectomy. The goal is to compare postoperative pain scores between patient groups receiving ESP block in lateral, prone, or sitting positions.

SECONDARY OUTCOMES:
Total Postoperative Analgesic Consumption | First 24 hours after surgery
  The cumulative dose (mg) of tramadol administered as rescue analgesia within the first 24 hours postoperatively will be recorded for each group.
Time to First Analgesic Request | Within 24 hours postoperatively
  The duration (in minutes) between the end of surgery and the patient's first request for additional analgesia.
Patient Satisfaction Score | 24 hours postoperatively
  Patient satisfaction will be assessed at 24 hours postoperatively using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied).
Skin-to-Target Distance | During preoperative ESP block procedure
  The distance (in millimeters) from the skin to the ESP block site will be measured via ultrasound at the T7 level in each patient position to determine anatomical variation.

CONTACTS AND LOCATIONS:
Overall Officials: Veli F Pehlivan, Asiss Prof, Principal Investigator — Harran University Faculty of Medicine, Department of Anesthesiology
Locations (1):
- Veli Fahri Pehlivan, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No